CLINICAL TRIAL: NCT06303869
Title: Deep Brain Stimulation Motor Ventral Thalamus (VOP/VIM) for Restoration of Speech and Upper-limb Function in People With Subcortical Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Gonzalez-Martinez (Other)
Responsible Party: Sponsor-Investigator, Jorge Gonzalez-Martinez, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY22070043
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Brain Disease; Central Nervous System Diseases; Nervous System Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Stroke; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Cardiovascular Diseases | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, open-label, descriptive, experimental.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Deep Brain Stimulation of the Motor Thalamus (Experimental): Individuals who have speech and motor deficits due to a stroke.
  Interventions: Device: Deep Brain Stimulation (DBS) of the Motor Thalamus

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) of the Motor Thalamus — All participants enrolled in this group will undergo a surgical procedure to implant deep brain stimulation electrode leads. The electrodes will be connected to external stimulators and a series of experiments will be performed to identify the types of movements that the hand and arm can make and how speech abilities are affected by the stimulation. The implant will be removed after less than 30 days.

SUMMARY:
The goal of this study is to verify whether the use of deep brain stimulation can improve motor function of the hand and arm and speech abilities for people following a stroke. Participants will undergo a surgical procedure to implant deep brain stimulation electrode leads. The electrodes will be connected to external stimulators and a series of experiments will be performed to identify the types of movements that the hand and arm can make and how speech abilities are affected by the stimulation. The implant will be removed after less than 30 days. Results of this study will provide the foundation for future studies evaluating the efficacy of a minimally-invasive neuro-technology that can be used in clinical neuro-rehabilitation programs to restore speech and upper limb motor functions in people with subcortical strokes, thereby increasing independence and quality of life.

DETAILED DESCRIPTION:
The study is designed to assess the assistive effects of DBS (i.e., immediate effects when the stimulation is turned ON) and obtain preliminary evidence for therapeutic effects (i.e., long-lasting effects with stimulation OFF). Researchers will 1) quantify the ability to recruit face muscles with electrical stimulation of the motor thalamus in patients with subcortical stroke, 2) quantify the ability to recruit arm and hand muscles with electrical stimulation of the motor thalamus in patients with subcortical stroke, and 3) verify if the delivery of DBS has effects on the central nervous system with clinical measures.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have suffered a single, ischemic, or hemorrhagic stroke more than 6 months before the time of enrollment with dysarthria as a result.
2. Participants must be between the ages of 18 and 75 years old. (Participants outside this age range may be at an increased medical risk and have an increased risk of fatigue during testing).
3. English speaker.
4. Participant must score ≤ 80% in at least 4 categories of the perceptual speech assessment (speech intelligibility, listener effort, speech naturalness, articulatory precision, speech rate, overall voice quality, and/or overall speech severity). OR ≤ 80% in at least 3 categories of the perceptual speech assessment AND ≤ 27 on the Communicative Participation Item Bank.

Exclusion Criteria:

1. Patients who refuse participation in the study.
2. Patients with gross anatomical variances in MR imaging or cerebral vascular accidents involving thalamic and cerebellar areas.
3. Patients with no clinical condition to undergo DBS implantation or highly dependent on anticoagulation therapy.
4. Patients who cannot undergo pre-operative MRIs or could not complete the pre-operative assessments.
5. Participants must not have any serious disease or disorder (ex. neurological condition other than stroke, cancer, severe cardiac or respiratory disease, renal failure, etc.) or cognitive impairments that could affect their ability to participate in this study.
6. Female participants of child-bearing age must not be pregnant, planning to become pregnant for the next 9 months, or breast feeding.
7. Participants must not be receiving anticoagulants.
8. Severe claustrophobia.
9. Participants must not be on anti-spasticity or anti-epileptic medications for the duration of the study.
10. Participants who have been deemed inappropriate for participation based upon results from the Brief Symptoms Inventory (BSI-18) and discussions with the Principal Investigator and a study physician
11. Evaluation to sign consent form score <12.
12. MRI contraindications (excluding subjects who are pregnant, who have metal in any portion of their body, have medical complications, cardiac pacemaker, cochlear implant, aneurysm clip, certain IUDs, or known problems of claustrophobia).
13. Medications with common cognitive side-effects.
14. Bleeding disorders or platelet dysfunction (e.g., from regular aspirin usage).
15. Patients must not have any lesions in the lower motoneuron causing flaccid dysarthria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 29 days
  The investigators will quantify the safety of DBS to treat post-stroke speech and upper-limb motor deficits. For this, the investigators will record all adverse events for the entire study duration. The study is considered successful if no serious adverse events related to the use of deep brain stimulation are reported.
Discomfort and Pain | Baseline, 2 weeks, 4 weeks, 6 months.
  The investigators will assess the relative level of discomfort and/or pain that is associated with the delivery of electrical stimulation to the motor thalamus. After each stimulation train patients will be asked to report a level of perceived discomfort using a 10 value subjective scale. Low values will be assigned to low discomfort and high values to high discomfort. The study is considered successful if 70% of recruited subjects do not report discomfort or pain at stimulation amplitudes that are required to obtain motor responses in the face and upper-limb muscles.

SECONDARY OUTCOMES:
Dysphagia | 29 days
  The investigators will use the modified barium swallow study (MBSS) to assess oropharyngeal swallow functions. This is a performance evaluation scale, that consist of 17 items with varying scales. The total score ranges from 0 to 55, where a higher score means a better outcome. Based on the preliminary data, the investigators will consider an increase of 1 point in at least 50% of the items of the Modified Barium Swallow Impairment Profile as a minimally acceptable improvement in swallow functions.
Hand dexterity | 29 days.
  The investigators will use the Box and Blocks Test to measure hand dexterity ability. Based on the preliminary data, the investigators will consider a percentage change of 18% as a minimally acceptable improvement in hand dexterity.
Muscle weakness | 29 days
  The investigators will measure muscle strength and range of motion produced by the subject during isometric facial movements (e.g. smile, tongue out, puckered lips, and open-close mouth). Based on the preliminary data, the investigators will consider an increase of 50% in ROM as a minimally acceptable improvement in muscle strength.
Dexterity of Articulation AMRs | 29 days
  The investigators will measure dexterity of articulation by alternating motion rates (AMRs) of the repetitive plosive sound (pah, tah, and kah). The investigators will consider an improvement of 10% in the rate to be minimally acceptable.
Dexterity of Articulation SMRs | 29 days
  The investigators will measure dexterity of articulation by sequential motion rates (SMRs) of the repetitive plosive sound (pah, tah, and kah). The investigators will consider an improvement of 10% in the rate to be minimally acceptable.
Intelligibility of Speech | 29 days
  The investigators will use the Assessment of Intelligibility of Dysarthric Speech (AIDS) to assess the quality of communication and intelligibility of speech at both word- and sentence-level. The investigators will consider an improvement of 5% correctly transcribed to be minimally acceptable.
Spasticity | 29 days
  Spastic dysarthria is characterized by a higher fundamental frequency (F0) of phoneme utterances than what is seen in normal speech. Thus, the investigators will quantify the degree of spasticity by calculating the F0 across a series of phonemes. The investigators will consider a reduction in F0 of 20% to be minimally acceptable.
Range of Motion (ROM) | 29 days
  The investigators will use the 2nd Edition Frenchay Dysarthria Assessment (FDA-2) to measure patterns of oral motor functions, with a particular focus on the following subsections: Respiration, Lips, Palate, Laryngeal, and Tongue. Each subsection is rated on a scale from "a" to "e", where "a" means normal for age, and "e" means unable to undertake task/movement/sound. So a score closer to "a" means a better outcome. The investigators will consider an improvement in severity level (e.g., from considerable to moderate severity, or a score of D to C) to be minimally acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gonzalez-Martinez, MD/PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with other researchers for the purpose of data analysis and collaboration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the end of the trial upon publication of the first manuscript. Estimation is 2 years from enrollment of the first participant.
Access Criteria: Data must be directly requested from the PI and will be shared upon completion of the necessary data-sharing agreement to protect confidential patient information.

REFERENCES:
- [Background] Ho, J. et al. TARGETED DEEP BRAIN STIMULATION OF THE MOTOR THALAMUS FACILITATES VOLUNTARY MOTOR CONTROL AFTER CORTICO-SPINAL LESIONS. medRxiv 2023-03 (2023).
- [Background] Lozano AM, Lipsman N, Bergman H, Brown P, Chabardes S, Chang JW, Matthews K, McIntyre CC, Schlaepfer TE, Schulder M, Temel Y, Volkmann J, Krauss JK. Deep brain stimulation: current challenges and future directions. Nat Rev Neurol. 2019 Mar;15(3):148-160. doi: 10.1038/s41582-018-0128-2. PMID 30683913
- [Background] Plow EB, Machado A. Invasive neurostimulation in stroke rehabilitation. Neurotherapeutics. 2014 Jul;11(3):572-82. doi: 10.1007/s13311-013-0245-y. PMID 24353109
- [Background] Molnar GF, Sailer A, Gunraj CA, Cunic DI, Lang AE, Lozano AM, Moro E, Chen R. Changes in cortical excitability with thalamic deep brain stimulation. Neurology. 2005 Jun 14;64(11):1913-9. doi: 10.1212/01.WNL.0000163985.89444.DD. PMID 15955943
- [Background] Baker KB, Plow EB, Nagel S, Rosenfeldt AB, Gopalakrishnan R, Clark C, Wyant A, Schroedel M, Ozinga J 4th, Davidson S, Hogue O, Floden D, Chen J, Ford PJ, Sankary L, Huang X, Cunningham DA, DiFilippo FP, Hu B, Jones SE, Bethoux F, Wolf SL, Chae J, Machado AG. Cerebellar deep brain stimulation for chronic post-stroke motor rehabilitation: a phase I trial. Nat Med. 2023 Sep;29(9):2366-2374. doi: 10.1038/s41591-023-02507-0. Epub 2023 Aug 14. PMID 37580534
- [Background] Cooper IS, Upton AR, Amin I. Reversibility of chronic neurologic deficits. Some effects of electrical stimulation of the thalamus and internal capsule in man. Appl Neurophysiol. 1980;43(3-5):244-58. doi: 10.1159/000102263. PMID 6975064
- [Background] Phillips NI, Bhakta BB. Affect of deep brain stimulation on limb paresis after stroke. Lancet. 2000 Jul 15;356(9225):222-3. doi: 10.1016/s0140-6736(00)02487-9. PMID 10963204
- [Background] Franzini A, Cordella R, Nazzi V, Broggi G. Long-term chronic stimulation of internal capsule in poststroke pain and spasticity. Case report, long-term results and review of the literature. Stereotact Funct Neurosurg. 2008;86(3):179-83. doi: 10.1159/000120431. Epub 2008 Mar 12. PMID 18334861